CLINICAL TRIAL: NCT04724850
Title: Observational Study About the Characteristics and Evolution of Patients Diagnosed With COVID-19 in Extremadura
Brief Title: Evolution of Coronavirus Disease 2019 (COVID-19) Patients in Extremadura
Acronym: COVIXTREM
Status: Completed | Type: Observational
Sponsor: Juan Fernando Masa Jiménez (Other)
Responsible Party: Sponsor-Investigator, Juan Fernando Masa Jiménez, Principal Investigator, University of Extremadura
Organization: University of Extremadura (Other)
Other Study IDs: 1/2020
Record Dates: First submitted 2021-01-11; First posted 2021-01-26 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Coronavirus Disease 2019
Keywords: Patients diagnosed with coronavirus disease 2019; Clinical characteristics of coronavirus disease 2019; Clinical evolution of coronavirus disease 2019; Effectiveness of drug treatment for coronavirus disease 2019
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Whole blood (only for prospectively recruited and consenting patients)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 patients: All patients diagnosed with COVID-19 in the community of Extremadura from the beginning of the epidemic to its ending in Spain.

SUMMARY:
At the end of January 2020, the international community was informed of the presence of a new viral disease that started in Wuhan (China) and spread rapidly throughout the world. The identified virus belonged to the coronavirus family (SARS-CoV-2) and the disease was named COVID-19. Today there are more than 2 million people diagnosed in Spain and more than 40 thousand in Extremadura. The partial knowledge about the development, evolution of the affected citizenship and their prognosis both early and late makes it necessary to analyze in depth their global and particular characteristics.

We will carry out a multicenter, observational, descriptive, cross-sectional and longitudinal study of patients diagnosed with SARS-CoV-2 virus infection in the Community of Extremadura to determine the effectiveness of drug treatments and the clinical and evolutionary characteristics of these patients and the different factors that may influence its evolution.

DETAILED DESCRIPTION:
Epidemiological, socio-sanitary, clinical, analytical and radiological data will be collected retrospectively and prospectively from all patients diagnosed with COVID-19 without hospital admission in our community from the start of the pandemic and for one year from the start of the study.

These data will be obtained mainly from the clinical history and collected in the data collection notebooks and electronic base designed for the study for subsequent analysis. The data collection period will be one year, estimating a sample of 5,000 patients.

In addition, patients included in the study prospectively will be asked for consent to collect a blood sample for freezing and storage in the Biobank of Extremadura and subsequent use to determine biomarkers and genetics.

The present study will be carried out in accordance with the observational National Post-Authorization Study (EPA) for medicines for human use proposed by Valdecilla Health Research Institute (IDIVAL), the main objective of which is to determine the effectiveness of the pharmacological treatments currently used in COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age and sex, including minors and pregnant women.
* Patients diagnosed with SARS-Cov2 infection according to the clinical and microbiological criteria established by the Health Authorities and clinical practice (these can be modified based on the Technical document "Clinical management of COVID-19" of the Ministry of Health) who require or not hospitalization and who receive or not specific pharmacologic treatment for the SARS-Cov2 infection.

Exclusion Criteria:

* Patients who do not give their informed consent to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with SARS-Cov2 infection according to the clinical and microbiological criteria established by the Health Authorities and clinical practice in the community of Extremadura in Spain, and who require or not hospitalization and who receive or not specific pharmacologic treatment for the SARS-Cov2 infection.
Sampling Method: Non-Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
To determine the effectiveness of the pharmacological treatments used for hospitalized patients with COVID-19 in clinical practice assessed in terms of mortality. | 28 days
  To determine the effectiveness of each drug the investigators will use the percentage of deceased subjects who were treated with each one of them.
To determine the effectiveness of the pharmacological treatments used in the clinical practice for hospitalized patients with SARS-Cov2 infection assessed by time until death. | 28 days
  To determine the effectiveness of each drug the investigators will use the time in days from the start to the pharmacological treatment to death.
To determine the effectiveness of the pharmacological treatments used in the clinical practice for hospitalized patients with SARS-Cov2 infection assessed in terms of recovery. | 28 days
  To determine the effectiveness of each drug the investigators will use the time from the start of the pharmacological treatment to recovery, understanding as recovery the disappearance of symptoms and two negative reverse transcription polymerase chain reaction (PCR) separated by at least 24 hours.

SECONDARY OUTCOMES:
To evaluate the influence of the age on the effectiveness of the pharmacological treatments used for hospitalized patients with SARS-Cov2 infection in clinical practice. | 28 days
  The investigators will analyze the effect of the age in years of the hospitalized patients on the effectiveness of the pharmacological treatments assessed in terms of mortality.
To evaluate the influence of the gender on the effectiveness of the pharmacological treatments used for hospitalized patients with SARS-Cov2 infection in clinical practice. | 28 days
  The investigators will analyze the effect of the gender (male or female) of the hospitalized patients on the effectiveness of the pharmacological treatments assessed in terms of mortality.
To evaluate the influence of the arterial hypertension on the effectiveness of the pharmacological treatments used for hospitalized patients with SARS-Cov2 infection in clinical practice. | 28 days
  The investigators will analyze the effect of the presence of arterial hypertension (yes or not) on the effectiveness of the pharmacological treatments in hospitalized patients assessed in terms of mortality.
To evaluate the influence of the diabetes on the effectiveness of the pharmacological treatments used for hospitalized patients with SARS-Cov2 infection in clinical practice. | 28 days
  We will analyze the effect of the presence of diabetes (yes or not) on the effectiveness of the pharmacological treatments in hospitalized patients assessed in terms of mortality.
To evaluate the influence of the dyslipidemia on the effectiveness of the pharmacological treatments used for hospitalized patients with SARS-Cov2 infection in clinical practice. | 28 days
  The investigators will analyze the effect of the presence of dyslipidemia (yes or not) on the effectiveness of the pharmacological treatments in hospitalized patients assessed in terms of mortality.
To evaluate the influence of myocardial infarction on the effectiveness of the pharmacological treatments used for hospitalized patients with SARS-Cov2 infection in clinical practice. | 28 days
  The investigators will analyze the effect of the presence of a history of myocardial infarction (yes or not) on the effectiveness of the pharmacological treatments in hospitalized patients assessed in terms of mortality.
To evaluate the influence of angina on the effectiveness of the pharmacological treatments used for hospitalized patients with SARS-Cov2 infection in clinical practice. | 28 days
  The investigators will analyze the effect of the presence of a history of angina (yes or not) on the effectiveness of the pharmacological treatments in hospitalized patients assessed in terms of mortality.
To evaluate the influence of chronic heart disease on the effectiveness of the pharmacological treatments used for hospitalized patients with SARS-Cov2 infection in clinical practice. | 28 days
  The investigators will analyze the effect of the presence of a history of chronic heart failure (yes or not) on the effectiveness of the pharmacological treatments in hospitalized patients assessed in terms of mortality.
To evaluate the influence of peripheral arterial disease the effectiveness of the pharmacological treatments used for hospitalized patients with SARS-Cov2 infection in clinical practice. | 28 days
  The investigators will analyze the effect of the presence of a history of peripheral arterial disease (yes or not) on the effectiveness of the pharmacological treatments in hospitalized patients assessed in terms of mortality.
To evaluate the influence of ictus on the effectiveness of the pharmacological treatments used for hospitalized patients with SARS-Cov2 infection in clinical practice. | 28 days
  The investigators will analyze the effect of the presence of a history of ictus (yes or not) on the effectiveness of the pharmacological treatments in hospitalized patients assessed in terms of mortality.
To influence of dementia on the effectiveness of the pharmacological treatments used for hospitalized patients with SARS-Cov2 infection in clinical practice. | 28 days
  The investigators will analyze the effect of the presence of a history of dementia (yes or not) on the effectiveness of the pharmacological treatments in hospitalized patients assessed in terms of mortality.
To evaluate the influence of neuromuscular disease on the effectiveness of the pharmacological treatments used for hospitalized patients with SARS-Cov2 infection in clinical practice. | 28 days
  The investigators will analyze the effect of the presence of a history of neuromuscular disease (yes or not) on the effectiveness of the pharmacological treatments in hospitalized patients assessed in terms of mortality.
To evaluate the influence of chronic obstructive pulmonary disease on the effectiveness of the pharmacological treatments used for hospitalized patients with SARS-Cov2 infection in clinical practice. | 28 days
  The investigators will analyze the effect of the presence of a history of chronic obstructive pulmonary disease (yes or not) on the effectiveness of the pharmacological treatments in hospitalized patients assessed in terms of mortality.
To evaluate the influence of asthma the effectiveness of the pharmacological treatments used for hospitalized patients with SARS-Cov2 infection in clinical practice. | 28 days
  The investigators will analyze the effect of the presence of a history of asthma (yes or not) on the effectiveness of the pharmacological treatments in hospitalized patients assessed in terms of mortality.
To evaluate de influence of chronic kidney disease the effectiveness of the pharmacological treatments used for hospitalized patients with SARS-Cov2 infection in clinical practice. | 28 days
  The investigators will analyze the effect of the presence of a history of chronic kidney disease (yes or not) on the effectiveness of the pharmacological treatments in hospitalized patients assessed in terms of mortality.
To evaluate the influence of the severity of the disease on the effectiveness of the pharmacologic treatments used for hospitalized patients with SARS-Cov2 infection in clinical practice assessed in terms of mortality. | 28 days
  To determine the severity of the disease, the investigators will use the following severity classification:
  Uncomplicated disease (symptoms of the upper respiratory tract with or without nonspecific symptoms: fever, muscle pain or atypical symptoms in the elderly), mild pneumonia (pneumonia confirmed on chest radiography and without signs of severity, with room air oxygen saturation > 90% and CURB65 score* ≤ 1), severe pneumonia (failure of > 1 organ or air ambient oxygen saturation < 90% or respiratory rate ≥ 30 rpm), respiratory distress (clinical findings, bilateral infiltrates on chest radiography and oxygenation deficit with PaO2 / FiO2 ≤ 300 mmHg), sepsis (organic dysfunction that can be identified as an acute change in the SOFA score > 2 points) and septic shock (arterial hypotension that persists after administration of resuscitation volume and that requires vasopressors to maintain a mean arterial pressure ≥ 65 mmHg and lactate ≥ 2 mmol / L in the absence of hypovolemia).
To evaluate the influence of taking non-steroidal anti-inflammatory drugs on the effectiveness of the pharmacological treatments used for SARS-Cov2 infection in hospitalized patients in clinical practice. | 28 days
  The investigators will analyze the effect of usual taking non-steroidal anti-inflammatory drugs (yes or not) on the effectiveness of the pharmacological treatments for SARS-Cov2 in hospitalized patients assessed in terms of mortality.
To evaluate the influence of taking angiotensin II receptor antagonists on the effectiveness of the pharmacological treatments used for SARS-Cov2 infection in hospitalized patients in clinical practice. | 28 days
  The investigators will analyze the effect of usual taking angiotensin II receptor antagonists (yes or not) on the effectiveness of the pharmacological treatments for SARS-Cov2 in hospitalized patients assessed in terms of mortality.
To evaluate the influence of taking oral anti-diabetics drugs on the effectiveness of the pharmacological treatments used for SARS-Cov2 infection in hospitalized patients in clinical practice. | 28 days
  The investigators will analyze the effect of usual taking oral anti-diabetics drugs (yes or not) on the effectiveness of the pharmacological treatments for SARS-Cov2 in hospitalized patients assessed in terms of mortality.
To evaluate the influence of administration of insulin on the effectiveness of the pharmacological treatments used for SARS-Cov2 infection in hospitalized patients in clinical practice. | 28 days
  The investigators will analyze the effect of usual administration of insulin (yes or not) on the effectiveness of the pharmacological treatments for SARS-Cov2 in hospitalized patients assessed in terms of mortality.
To obtain information on the dosage of the pharmacologic treatments used for the treatment of the SARS-Cov2 infection in hospitalized patients and outpatients in clinical practice. | During the drug treatment, an average of two weeks
  The investigators will collect the dosage of each drug used in clinical practice (amount of drug administered, usually in milligrams, per time interval in hours)
To obtain information on the duration of the pharmacologic treatments used for the treatment of the SARS-Cov2 infection in hospitalized patients and outpatients in clinical practice. | During the drug treatment, an average of two weeks
  The investigators will collect the days of use of each drug.
To identify and quantity the side effects of the pharmacologic treatments used for the treatment of the SARS-Cov2 infection in hospitalized patients and outpatients in clinical practice. | 3 months
  The investigators will collect any side effect, the suspected causative drug, start and end data of the side effect, if it is severe or not and the outcome (full recovery, recovery with sequelae or death).
To analyze the effectiveness of the pharmacologic treatments used for SARS-Cov2 infection in hospitalized patients in clinical practice assessed by time of hospitalization. | 180 days
  The investigators will use the hospitalization days of the patients treated with each drug used for the treatment of SARS-Cov2.
To analyze the effectiveness of the pharmacologic treatments used for SARS-Cov2 infection in hospitalized patients in clinical practice assessed by the need to stay in the intensive care unit. | 28 days
  The investigators will analyze the percentage of patients treated with each drug that need admission to the intensive care unit and the mean number of days that they remained in that unit.
To analyze the effectiveness of the pharmacologic treatments used for SARS-Cov2 infection in hospitalized patients in clinical practice assessed by the maximum severity reached during admission. | 28 days
  To determine the maximum level of severity reached, the investigators will use the following classification:
  Uncomplicated disease (symptoms of the upper respiratory tract with or without nonspecific symptoms), mild pneumonia (confirmed on chest radiography and without signs of severity, with room air oxygen saturation > 90% and Pneumonia Severity Score (CURB65) ≤ 1), severe pneumonia (failure of > 1 organ or air ambient oxygen saturation < 90% or respiratory rate ≥ 30 rpm), respiratory distress (bilateral infiltrates on chest radiography and oxygenation deficit with partial pressure of oxygen / inspiratory oxygen fraction ≤ 300 mmHg), sepsis (organic dysfunction with an acute change in the Sequential Organ Failure Assessment Score > 2 points) and septic shock (arterial hypotension that persists after administration of resuscitation volume and that requires vasopressors to maintain a mean arterial pressure ≥ 65 mmHg and lactate ≥ 2 mmol / L in the absence of hypovolemia)
To determine the evolution of patients with a positive diagnostic test for SARS-Cov2 who have not been treated with some of the specific drugs for this disease used for hospitalized patients in clinical practice. | 28 days
  To determine the evolution of this group of patient the investigators will use the need admission on the intensive care unit or respiratory intermediate care unit, the need of ventilatory support (conventional oxygen therapy, high-flow oxygen therapy, invasive or non-invasive ventilation, prone position, extracorporeal membrane oxygenation), recovery or death and medical complications during admission (other infections, severe arrhythmia, respiratory distress, kidney failure, heart failure, myocardial infarction, angina, auricular fibrillation / flutter, stroke and others).
To describe the symptoms presented by the hospitalized patient for COVID-19 in the Community of Extremadura during the entire epidemic period | 7 days
  The investigators will collect the presence of the main symptoms on admission: fever, shaking chills, cough, expectoration, hemoptysis, dyspnea, chest pain, headache, diarrhea, asthenia, anorexia, malaise, anosmia, dysgeusia, nasal obstruction, rhinorrhea, odynophagia, myalgia or body pain, weight loss, nausea and vomiting
To describe the temperature presented during admission by patients hospitalized for COVID-19 in the community of Extremadura during the entire period of the pandemic. | 28 days
  The investigators will collect the temperature in degrees centigrade on admission and every seven days during admission
To describe the heart rate presented during admission by patients hospitalized for COVID-19 in the community of Extremadura during the entire period of the pandemic. | 28 days
  The investigators will collect the heart rate in beats per minute on admission and every seven days during admission.
To describe the oxygen saturation breathing ambient air presented during admission by patients hospitalized for COVID-19 in the community of Extremadura during the entire period of the pandemic. | 28 days
  The investigators will collect the oxygen saturation breathing ambient air by arterial blood gases or pulse oximetry, depending on availability, on admission and every seven days during admission.
To describe the blood pressure presented during admission by patients hospitalized for COVID-19 in the community of Extremadura during the entire period of the pandemic. | 28 days
  The investigators will collect the blood pressure in millimeters of mercury on admission and every seven days during admission.
To describe the symptoms presented by the outpatients diagnosed with COVID-19 in the Community of Extremadura during the entire epidemic period. | 28 days
  The investigators will collect the presence of the main symptoms during the follow-up: fever, shaking chills, cough, expectoration, hemoptysis, dyspnea, chest pain, headache, diarrhea, asthenia, anorexia, malaise, anosmia, dysgeusia, nasal obstruction, rhinorrhea, odynophagia, myalgia or body pain, weight loss, nausea and vomiting on diagnosis and every seven days during de follow up.
To describe the temperature presented by the outpatients diagnosed with COVID-19 in the Community of Extremadura during the entire epidemic period. | 7 days
  The investigators will collect the temperature in degrees centigrade at diagnosis.
To describe heart rate presented by the outpatients diagnosed with COVID-19 in the Community of Extremadura during the entire epidemic period. | 7 days
  The investigators will collect the heart rate in beats per minute at diagnosis.
To describe the respiratory rate presented by the outpatients diagnosed with COVID-19 in the Community of Extremadura during the entire epidemic period. | 7 days
  The investigators will collect the respiratory rate in breaths per minute at diagnosis
To describe the oxygen saturation breathing ambient air presented by the outpatients diagnosed with COVID-19 in the Community of Extremadura during the entire epidemic period. | 7 days
  The investigators will collect the oxygen saturation breathing ambient air by arterial blood gases or pulse oximetry, depending on availability, at diagnosis.
To describe the blood pressure presented by the outpatients diagnosed with COVID-19 in the Community of Extremadura during the entire epidemic period. | 7 days
  The investigators will collect the blood pressure in millimeters of mercury at diagnosis.
To describe the radiological findings in hospitalized patients with CIVID-19 in the Community of Extremadura during the entire epidemic period. | 28 days
  The investigators will collect the radiological findings of the chest radiograph and the computed tomography (CT) according to two classifications:
  Unilateral or bilateral alveolar infiltrate, diffuse intersticial infiltrate, pattern on ground glass, pleural effusion and normal.
  Intersticial infiltrate, lobar or bilobar alveolar infiltrate, unilateral or bilateral alveolar lung infiltrate with three degrees of severity (mild, moderate or severe with <25%, 25-50% or >50% of lung affected, respectively), pleural effusion and normal.
  These findings will be collected weekly during admission to the conventional ward and daily during admission to intensive or intermediate respiratory care unit.
To describe the radiological findings in outpatients with CIVID-19 in the Community of Extremadura during the entire epidemic period. | 7 days
  The investigators will collect the radiological findings of the chest radiograph and the computed tomography (CT) according to two classifications:
  Unilateral or bilateral alveolar infiltrate, diffuse intersticial infiltrate, pattern on ground glass, pleural effusion and normal.
  Intersticial infiltrate, lobar or bilobar alveolar infiltrate, unilateral or bilateral alveolar lung infiltrate with three degrees of severity (mild, moderate or severe with <25%, 25-50% or >50% of lung affected, respectively), pleural effusion and normal.
  These findings will be collected at diagnosis.
To describe the ferritin levels in the blood of hospitalized patients with COVID-19 in the Community of Extremadura during the entire epidemic period. | 28 days
  The investigators will collect the ferritin levels in nanogram per milliliter, weekly during admission to the conventional ward and daily during admission to intensive or intermediate respiratory care unit.
To describe the D-dimer levels in the blood of hospitalized patients with COVID-19 in the Community of Extremadura during the entire epidemic period. | 28 days
  The investigators will collect the D-dimer levels in nanogram per milliliter, weekly during admission to the conventional ward and daily during admission to intensive or intermediate respiratory care unit.
To describe the interleukin 6 levels in the blood of hospitalized patients with COVID-19 in the Community of Extremadura during the entire epidemic period. | 28 days
  The investigators will collect the interleukin 6 levels in picogram per milliliter, weekly during admission to the conventional ward and daily during admission to intensive or intermediate respiratory care unit
To describe the lymphocyte count in the blood of hospitalized patients with COVID-19 in the Community of Extremadura during the entire epidemic period. | 28 days
  The investigators will collect the lymphocyte count expressed in 10*3 per milliliter, weekly during admission to the conventional ward and daily during admission to intensive or intermediate respiratory care unit
To describe the c-reactive protein level in the blood of hospitalized patients with COVID-19 in the Community of Extremadura during the entire epidemic period. | 28 days
  The investigators will collect the c-reactive protein level in milligrams per deciliters, weekly during admission to the conventional ward and daily during admission to intensive or intermediate respiratory care unit.
To describe the results of SARS-CoV2 diagnostic test performed in hospitalized patients with COVID-19 in the Community of Extremadura during the entire epidemic period. | 21 days
  The investigators will collect the result (positive or negative) of all tests performed to confirm the diagnosis of SARS-CoV2 infection: polymerase chain reaction test, serological test and antigen detection test.
To describe the ferritin levels in the blood of outpatients with COVID-19 in the Community of Extremadura during the entire epidemic period. | 7 days
  The investigators will collect the ferritin levels in nanogram per milliliter at diagnosis.
To describe the D-dimer levels in the blood of outpatients with COVID-19 in the Community of Extremadura during the entire epidemic period. | 7 days
  The investigators will collect the D-dimer levels in nanogram per milliliter at diangosis.
To describe the interleukin 6 levels in the blood of outpatients with COVID-19 in the Community of Extremadura during the entire epidemic period. | 7 days
  The investigators will collect the interleukin 6 levels in picogram per milliliter at diagnosis.
To describe the lymphocyte count in the blood of outpatients with COVID-19 in the Community of Extremadura during the entire epidemic period. | 7 days
  The investigators will collect the lymphocyte count expressed in 10*3 per milliliter diagnosis.
To describe the c-reactive protein level in the blood of outpatients with COVID-19 in the Community of Extremadura during the entire epidemic period. | 7 days
  The investigators will collect the c-reactive protein level in milligrams per deciliters at diagnosis.
To describe the results of SARS-CoV2 diagnostic test performed in outpatients with COVID-19 in the Community of Extremadura during the entire epidemic period. | 14 days
  The investigators will collect the result (positive or negative) of all tests performed to confirm the diagnosis of SARS-CoV2 infection: polymerase chain reaction test, serological test and antigen detection test.
To assess the health-related quality of life perceived by hospitalized patients after recovery. | Up to six months
  To determine the quality of life related to health the investigators will use the Short Form-12 Health Survey after recovery. This questionnaire assesses the degree of well-being and functional capacity and it is composed of twelve items and eight dimensions (physical function, physical role, body pain, mental health, general health, vitality, social function and emotional role), defining a positive or negative state of the physical and mental health. Some included items are: "In general, would you say that your health is", "During the last 4 weeks, to what extent has your physical health or emotional problems hindered your usual social activities with family, friends, neighbors or other people? "," Did you have pain in any part of your body during the last 4 weeks? ". The response options form Likert-type scales where the number of options varies from three to six points. The score ranges from 0 to 100. A higher score implies a better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Juan F Masa Jiménez, PhD, Principal Investigator — Servicio Extremeño de Salud
Locations (1):
- Hospital San Pedro de Alcántara, Cáceres, Spain

IPD SHARING:
Plan to Share IPD: Yes
Additional related documents such as study protocol, statistical analysis plan and informed consent form will be available upon request from the project principal investigator.
  (Dr. Juan Fernando Masa Jiménez). De-identified patients´data can be requested by researchers for use in independent scientific research and will provided following review and approval of the research proposal (including statistical analysis plan) and completion of a data sharing agreement with the Project Publications Committee. Investigator Data requests can be made anytime from 1 to 2 years after the publication of this trial. Requests should be sent to the corresponding author (Dr. Juan Fernando Masa Jiménez- fmasa@separ.es)